CLINICAL TRIAL: NCT02968680
Title: Pilot Translational Study of Sonazoid-Enhanced Ultrasonography for Sentinel Lymph Node Mapping in Cutaneous Melanoma
Brief Title: Sonazoid-Enhanced Ultrasound in Detecting Sentinel Lymph Node in Patients With Cutaneous Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10M-15-3; NCI-2016-01088 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10M-15-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-08-02; First posted 2016-11-18 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Cutaneous Melanoma; Melanoma
MeSH Terms: conditions — Melanoma | interventions — Sentinel Lymph Node Biopsy; Ultrasonography; Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (sonazoid, ultrasound imaging, SLNB) (Experimental): Patients receive sonazoid ID and undergo ultrasound imaging. Patients also undergo standard of care SLNB.
  Interventions: Procedure: Sentinel Lymph Node Biopsy; Device: Ultrasonography; Drug: Sonazoid

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy — Undergo SLNB
  Other Names: Sentinel Node Biopsy; Sentinel node biopsy alone; SLNB; SNB
Device: Ultrasonography — Undergo sonazoid-enhanced ultrasonography
  Other Names: ULTRASOUND; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US
Drug: Sonazoid — Patients receive sonazoid intradermally (ID) and undergo ultrasound imaging.
  Other Names: Contrast ultrasound microvascular perfusion imaging

SUMMARY:
This pilot phase I trial studies how well sonazoid-enhanced ultrasound works in detecting sentinel lymph node in patients with cutaneous melanoma. Sonazoid is a contrast agent that may make it easier to see if the tumor cells have spread to the sentinel lymph node using an ultrasound.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study the imaging feasibility of peri-tumoral administration of sonazoid ultrasound contrast agent for assessment of sentinel lymph node (SLN) detection in melanoma.

II. To compare SLN detection between sonazoid ultrasound and standard of care (SOC) technique.

SECONDARY OBJECTIVES:

I. To assess the sonazoid ultrasound (US) imaging appearance of lymph nodes which are shown to be involved with metastatic disease.

OUTLINE:

Patients receive sonazoid intradermally (ID) and undergo ultrasound imaging. Patients also undergo standard of care sentinel lymph node biopsy (SLNB).

After completion of study treatment, patients are followed up at 24 and 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous melanoma with Breslow depth > 1 mm or melanoma Breslow depth of 0.76 - 1.00 mm in setting of ulceration, extensive regression
* Mitotic rate >= 1/mm^2
* Presence of angiolymphatic invasion
* Deep positive margin
* No known allergies to contrast material

Exclusion Criteria:

* Pregnant or nursing
* Patients with known cardiac shunt
* Patients with class II heart failure or worse, per New York Heart Association (NYHA) classification
* Patients who have experienced an acute coronary syndrome or angina in the past 6 months
* Patients who have undergone coronary artery bypass grafting (CABG) or coronary stenting in the past 3 years
* Patients with evidence of moderate or severe cardiac valvular disease on echocardiogram
* Patients with evidence of moderate or severe pulmonary hypertension on echocardiogram
* Patients with stage II chronic obstructive pulmonary disease (COPD) or worse, per Global Initiative for Chronic Obstructive Lung Disease (GOLD) classification
* Patients with hypersensitivity to sonazoid or one of its components
* Patients with hypersensitivity to egg or egg products, because sonazoid contains a chicken egg-derived surfactant (hydrogenated egg phosphatidylserine sodium)
* Patients who cannot consent for themselves

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Percent of patients with SLN identified by sonazoid-US alone or both sonazoid-US and conventional methods | Up to 1 year
  Analyzed using descriptive comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin King, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States